CLINICAL TRIAL: NCT03346486
Title: Open, Fixed Sequence Diet-switch 4-week Intervention on the Effects of Brain-friendly Diet on Metabolic and Physiological Parameters and Cognitive Performance in Office Workers at Assumed Metabolic Risk
Brief Title: Dietary Intervention With Brain-friendly Diet
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fazer Group (Industry)
Collaborators: Nokia Technologies Oy (Unknown); Nightingale Health Oy (Unknown); Tekes - the Finnish Funding Agency for Innovation (Unknown); Finnish Institute of Occupational Health (FIOH) (Unknown); Oy Medfiles Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MFBF008 BRAVE
Record Dates: First submitted 2017-08-24; First posted 2017-11-17 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2017-09

CONDITIONS: Physiological Stress; Cognitive Performance; LDL Cholesterol
Keywords: Diet; Metabolites; Cognitive function; Physiology; LDL; Diet Habit; Diet Modification
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Open, fixed sequence diet-switch 4-week intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control diet (Placebo Comparator): Regular diet
  Interventions: Other: Control diet
- Intervention diet (Active Comparator): Brainfood diet
  Interventions: Other: Intervention diet

INTERVENTIONS:
Other: Control diet — Regular diet
  Arms: Control diet
Other: Intervention diet — Brainfood dietary regime planned to be optimal for metabolism and cognitive function; having focus on regular meal frequency (breakfast, lunch and afternoon snack) and well-balanced light lunch at work according to the so-called plate model and optimized recipes- will be provided.
  Other Names: Brainfood diet
  Arms: Intervention diet

SUMMARY:
To evaluate the effect of dietary intervention on metabolic risk profile, and on potential simultaneous changes in physiological and cognitive functions and to collect a unique database using state-of-the-art technologies on variables related to the above mentioned areas.

DETAILED DESCRIPTION:
The study is compiled from 4 phases: 1) a pilot study to evaluate performance and feasibility of the measurements and logistics for the BRAVE intervention study (N=10), 2) a pre-screening phase to select volunteers for the intervention study based on metabolite analyses (N=600), 3) the BRAVE intervention study as a controlled non-randomized open-label fixed sequence diet switch trial (N=88)and 4) a non-interventional reference group to estimate the learning effect due to repeated cognitive testing (N=30).

The Brainfood dietary regime is planned optimal for metabolism and cognitive function; having focus on regular meal frequency (breakfast, lunch and afternoon snack) and well-balanced light lunch at work -according to the so-called plate model and optimized recipes- will be provided.

ELIGIBILITY:
Inclusion criteria

1. Signed written informed consent
2. Age 18-65 years
3. Assumed metabolic risk based on pre-screening assessment of glucose and lipid metabolism related metabolites defined initially as being within the most impaired quartile with reference to available metabolite data-base from a comparable population. If recruitment efficiency requires, having a metabolic profile within the most impaired half instead of a quartile may be applied.
4. Male or female with at least 1/3 of the gender defined predominant among screened participants with assumed metabolic risk
5. Adequate Finnish or English skill to comprehend trial related instructions and questionnaires
6. Chest circumference of 75 to 115 cm (limits included)

Exclusion criteria

1. High probability to travel for more than one working day a week during the trial
2. Expected or planned major changes in lifestyle (diet, level of exercise, significant changes in work) or involved in the R&D of the measuring devices applied in the trial
3. Allergies restricting compliance with control or intervention diet (celiac disease, gluten free diet, stringent FODMAP diet)
4. Nickel allergy
5. History of unstable coronary artery disease (myocardial infarction, coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA), temporal ischemic attack within the previous 6 months
6. Diagnosed type 1 or type 2 diabetes requiring treatment
7. Inflammatory bowel disease or other intestinal or oesophageal disease requiring medical treatment or likely to have a nutritional affect
8. History of malignant diseases like cancer within five years prior to recruitment
9. Lipid lowering medication (statin, cholestyramine) or medication for obesity (orlistat, or liraglutide) or depression
10. Alcohol abuse (> 4 portion/per day) or recreational drug abuse
11. Pregnancy or planned pregnancy or lactating
12. Suspected low compliance according to the investigator's assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Change in LDL cholesterol | 8 weeks
  Change in serum LDL concentration between control period and intervention period

SECONDARY OUTCOMES:
Change in serum metabolite concentrations | 8 weeks
  Change in serum metabolite concentrations
Change in cognitive performance | 4 weeks
  Change in cognitive performance
Changes in self-reported vigilance | 4 weeks
  Changes in self-reported vigilance
Changes in self-reported task load | 4 weeks
  Changes in self-reported task load
Daily pulse profile (evening- night- morning) | 8 weeks
  Changes in pulse profile (evening- night- morning), mean level, between control period and intervention period
Daily profile of heart rate variability (evening- night- morning) | 8 weeks
  Changes in heart rate variability profile (evening- night- morning), between control period and intervention period
Change in dietary habits and nutrient intake | 8 weeks
  Change in dietary habits and nutrient intake according to a standard 3-day food record between control period and intervention period
Number of adverse events | 8 weeks
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Arja Uusitalo, MD, Principal Investigator — FIOH
Locations (1):
- Medfiles BRAVE clinic, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No